Assessing and Enhancing Emotional Competence for Well-Being (ECoWeB) in Young Adults: A principled, evidence-based, mobile-health approach to prevent mental disorders and promote mental well-being



Trial Consent forms A and B Version 1.0 dated 10.09.2020

Consent Form A- Consent for Assessment (Online Format)

Consent Form B- Consent to enter the Trial (Online Format)



## **CONSENT FORM A**

Title of Project: Assessing and Enhancing Emotional Competence for Well-Being (ECoWeB) in the Young:

Consent A

| | | | | Please<br>Tick box |
|---|---|---|---|---|
| 1) I understand that I am consenting to complete online questionnaires and tasks to check if tapart in the ECoWeB study is right for me. | | | | |
| 2) I understand that all my data will be kept confidential and stored securely. My contact details will be kept separately from other information. My contact details will be permanently deleted by the end of September 2022 (anticipated study end). My other data will be kept for 7 years for research purposes only. This is in line with good research practice. | | | | |
| | | voluntary. I am free to v<br>deleted at any time until | vithdraw at any time without<br>the study ends. | giving |
| 4) I understand that the data collected from me (without my contact details) will be shared with researchers and collaborators within the EcoWeb Consortium. | | | | |
| 5) I am aged between 16 years and 22 years old. | | | | |
| 6) I confirm that I have read the information sheet dated 10.09.2020 (version 0.9) for the above study. I have been provided with a phone number and email address so that I can ask any questions. | | | | |
| 7) I agree to take part i<br>I will be informed that | | | understand that it is possible | |
| Name of Participant | Date | | Signature | |
| Autocomplete | | | | |
| Name of Person | Date | Signature | taking consent | |
| Email address | | Phone number | | |

The consent form and info sheet are now automatically sent to the ppt by email after completion and before this point.



| Centre: | Participant Identification Number for this trial: |
|---|---|
| CONSENT FORM B | |
| Title of Project: <b>Assessing and Enh Young</b> | ancing Emotional Competence for Well-Being (ECoWeB) in the |
| Consent B | |
| | Please tick box |
| 1) I consent to take part in this res<br>test the benefits of different Apps | earch about emotion and well-being in young people which will for mental well-being. |
| wellbeing over one year at three for | in the study I will be assessed on my emotional experiences and ollow up web-based assessments. I will also use the Smartphone ne App for a month. I commit to completing these assessments. |
| • | als will be selected at random (by chance) to be offered additional to improve emotional skills and well-being versus not being |
| • | udy does not replace any medical treatment/help I may need. My or my medical care. I will contact them should I feel at risk to |
| - | study only offers self-monitoring and self-help. It does not provide I nor directly supported by clinicians or therapists. I understand lelp if I feel distressed or at risk. |
| be kept separately from other data<br>deleted by the end of September 2 | rill be kept confidential and stored securely. My contact details will a collected on the website and the App. My contact details will be 2022 (anticipated study end). My other data will be kept for 7 This is in line with good research practice. |
| 7) I understand that my participati any reason. | on is voluntary. I am free to withdraw at any time without giving |
| I can voluntarily choose to vocally passive recording at any time. I un then put together again in a rando my identity. These reordered voice | n Diary in the App, I can take part in research into voice and mood. record an emotional event or not each time. There will be no derstand that each recording will be broken up into tiny bits and om order. This means that no-one can hear what I said and hides e files will be automatically analysed on the App to identify encrypted and sent to a secure server for further analysis. The app mood states in my voice. |
| | y record emotional events, then the content-free voice files and e consortium for research into mood and voice. |
| 10) I understand that all my data v<br>stored safely on a password protect | vill be encrypted before transfer between research partners and cted server. |
| 11) I understand that I can ask for unless it is no longer connected to | any of my data (including voice files) to be deleted at any time my contact details. |

| 12) I understand that data collected from me will be shared with researchers and collaborators within the EcoWeb Consortium and may be used to support other research in the future. | | | |
|---|---|---|---|
| 12\ I confirm that I have | a had the ennertunity ! | o road the infor | mation in Varsian 0.0 of the |
| 13) I confirm that I have had the opportunity to read the information in Version 0.9 of the information sheet dated 10.09.2020. I have had the opportunity to ask any questions I have. These | | | |
| questions were answered satisfactorily. The information sheet provides contact details for the | | | |
| researchers in my country for any future questions I might have. | | | |
| 14) I confirm that I am aged between 16 years and 22 years old. | | | |
| ACVI - Idella ta la construit de la construit | | | |
| 15) I would like to be contacted about opportunities to take part in additional collaborative research with researchers from the University of Oxford (optional) | | | |
| 16) Based on the above, I agree to take part in the ECoWeb study. | | | |
| 10) based on the above, ragree to take part in the Ecover Study. | | | |
| Name of Participant | Date | | Signature |
| Autocomplete | | | |
| Name of Person | Date | Signature | taking consent |
| to call. This can be a re | lative, guardian, doctor | or long-term fr | i, we would like to have someone else iend who knows you well and is over re very concerned about you and could |
| Trusted person contact details- Name | | ph | phone number |